CLINICAL TRIAL: NCT06563154
Title: Investigation of the Relationship Between Exercise Capacity, Physical Fitness, Quality of Life, Physical Activity Level, Cognitive Status and Health Literacy in Individuals Diagnosed With Dyslipidemia
Brief Title: Are Exercise Capacity and Physical Fitness Related With Quality of Life, Physical Activity, Cognitive Health and Health Literacy in Dyslipidemia
Status: Completed | Type: Observational
Sponsor: Çankırı Karatekin University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Furkan Özdemir, Lecturer, Çankırı Karatekin University
Other Study IDs: 03-01-2023-4
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemia; Exercise Capacity; Physical Fitness; Cognitive Health; Physical Activity; Health Literacy
MeSH Terms: conditions — Dyslipidemias; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Group
  Interventions: Diagnostic Test: Exercise Capacity Assessment; Diagnostic Test: Physical Fitness Assessment; Other: Quality of Life Assessment; Other: Physical Activity Assessment; Other: Cognitive Health Assessment; Other: Health Literacy Assessment

INTERVENTIONS:
Diagnostic Test: Exercise Capacity Assessment — To examine the relationship between exercise capacity and physical fitness of dyslipidemia patients and quality of life, cognitive status and health literacy.
Diagnostic Test: Physical Fitness Assessment — * 1-Minute Sit-to-Stand Test: Participants will be asked to sit down and stand up for 1 minute without pausing, and the repetition number will be recorded.
  * Timed Up-and-Go Test: Participants will be asked to get up, walk a distance of 3 meters, return and sit down again. The time spent during this track will be recorded.
  * Peripheral muscle strength assessment: Participants will be asked to resist the resistance by producing maximum isometric force during the movement, and the maximal force will be evaluated with a dynamometer. The quadriceps femoris muscle, shoulder abductor muscles and hand grip strength will be used for the assessment.
  * Flexibility assessment: Participants will be asked to reach towards the tips of their toes while sitting. During this time, the distance between the participant's fingertips and toes will be measured.
Other: Quality of Life Assessment — Participants' quality of life will be assessed with the Turkish version of the Short Form Quality of Life Questionnaire (SF-36). The questionnaire consists of 36 questions that examine quality of life from different perspectives. It examines quality of life in the subcategories of physical function, physical role difficulty, pain, general health, vitality (energy), social function, emotional role difficulty and mental health. The score for each category varies between 0-100, with a high score indicating a good quality of life.
Other: Physical Activity Assessment — Participants' physical activity level will be assessed with the Turkish version of the International Physical Activity Scale - Short Form (IPAQ-SF). The IPAQ-SF evaluates the physical activities of the participants in the last 7 days based on sitting time, walking time, moderate and vigorous physical activities.
Other: Cognitive Health Assessment — Participants' cognitive health will be assessed with the with the Turkish version of the Mini Mental State Examine (MMSE). The test is scored between 0-30. Scores of 25 and above are considered normal. A total score of less than 10 indicates severe impairment. Scores between 10-19 indicate moderate dementia. Scores between 19-24 indicate early dementia.
Other: Health Literacy Assessment — Participants' health literacy will be assessed with the Turkish version of the HLS-EU-47 health literacy survey. The survey consists of 47 questions. Each item is assessed with one of the following options: Very difficult (1), difficult (2), easy (3), very easy (4) and I don't know. A high total score indicates good health literacy. A total score of 0-25 points indicates insufficient health literacy, >25-33: problematic - limited health literacy, >33-42: sufficient health literacy, >42-50: excellent health literacy.

SUMMARY:
There is insufficient literature explaining the relationship between exercise capacity and physical fitness of dyslipidemia patients and quality of life, cognitive status and health literacy. Our aim with this study is to provide more information to the scientific literature about the relationship between exercise capacity and physical fitness and quality of life and health literacy in dyslipidemia patients.

DETAILED DESCRIPTION:
Lipid profile disorders (especially high total blood cholesterol levels) are considered a significant public health problem worldwide and it is reported that approximately one in three people are exposed to risk factors that can lead to dyslipidemia. Prevalence studies conducted worldwide show that lipid profile disorders vary between 6.9% and 43.6%. Today, ischemic heart and central nervous system diseases are reported to be the most important causes of mortality and morbidity in the adult population globally. It is accepted that lipid profile disorders are the leading risk factors that cause ischemic heart diseases in particular. Since lipid profile disorders are caused by many different genetic and environmental factors, their incidence varies according to regions, lifestyle habits and individual factors. Apart from individual factors, lipid weight in the diet and lack of other nutrients that balance lipid metabolism, physical activity level and inactivity, other existing comorbid diseases and medical treatments change lipid metabolism in individuals and may lead to deterioration in lipid profile. In particular, lifestyle habits are the most easily modifiable factors that affect lipid metabolism. Studies conducted to evaluate the effect of genetic factors have shown that blood lipid levels are generally higher in Caucasians (especially total plasma cholesterol), that plasma high-density lipoprotein (HDL) levels are lower in East-Southeast Asian societies, and that plasma lipid density is generally lower in Hispanic societies. These studies have also indicated that these differences in lipid profiles are seen in the ethnic group examined in isolation when compared to other ethnic groups living in the same region, and therefore that dyslipidemia also has a genetic origin. It is recommended to follow multifaceted approaches when treating lipid profile disorders. Dietary counseling and exercise therapy are generally recommended to be included in these approaches. Exercise therapy is considered a very important treatment option, especially for controlling and treating obesity, hypertension, hyperglycemia, and metabolic syndrome symptoms that may accompany dyslipidemia. Physical activity is defined as body movements that create skeletal muscle contraction and increase energy expenditure. Exercise is a specialized type of physical activity that focuses on working specific muscle groups within a structured program for a specific purpose. Physical activity and exercise are beneficial for health and have a positive effect on psychological function, quality of life, morbidity, and cardiorespiratory fitness. Physical activity and exercise also increase self-esteem and social participation, while reducing depression and other related mental symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Being followed up with a diagnosis of dyslipidemia,
* Being between the ages of 18-65,
* Being willing to participate in the study.

Exclusion Criteria:

* Having an orthopedic, neurological, cardiac, pulmonary or rheumatological disease that may affect functional capacity,
* Having a psychiatric disorder that may affect cooperation,
* Refusing to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dyslipidemia
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | First Day
Physical Fitness | Second Day

SECONDARY OUTCOMES:
Physical Activity | Second Day
Quality of Life Assessment | Second Day
Cognitive Health | Second Day
Health Literacy | Second Day

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozdemir F, Saglam M, Uyaroglu OA, Vardar Yagli N. Impact of physical activity, health literacy and cognitive health on quality of life in dyslipidemia: an observational study. Sci Rep. 2025 Oct 13;15(1):35586. doi: 10.1038/s41598-025-02223-4. PMID 41083504